CLINICAL TRIAL: NCT02205502
Title: Efficacy of Lidocaine as Local Anesthetics in Children Under Procedural Sedation and Analgesia Using Ketamine
Brief Title: Lidocaine as Local Anesthetics in Children Under Ketamine Sedation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin Hee Lee, Assistant Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Lidocaine-01
Record Dates: First submitted 2014-06-16; First posted 2014-07-31 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Conscious Sedation Failure During Procedure; Analgesia; Anesthesia
MeSH Terms: conditions — Agnosia | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine (Experimental): Proper amount of lidocaine will be injected lacerated wound.
  * dosage form: fluid
  * dosage: not exceeding 1mg/kg
  * frequency: once
  * duration: n/a
  Interventions: Drug: Lidocaine
- Normal saline (Placebo Comparator): Normal saline will be used as a placebo for lidocaine
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Lidocaine — Normal saline will be injected subcutaneously as a placebo for lidocaine in study group of children.
  Arms: Lidocaine
Drug: Normal saline
  Arms: Normal saline

SUMMARY:
Ketamine seems an obvious choice in the setting of an emergency department in laceration repair.

Lidocaine is the local anesthetics widespread used.

Ketamine leads to dissociative amnesia.

Theoretically , lidocaine is not useful in laceration repair using ketamine.

However, lidocaine is used with ketamine in many emergency department.

The investigators compare lidocaine with placebo as an adjunct to ketamine sedation in children undergoing primary closure

ELIGIBILITY:
Inclusion Criteria:

* patients who need suturing for laceration under procedural anesthesia using ketamine

Exclusion Criteria:

* contraindication to ketamine and lidocaine
* patients involved to other studies
* more or equal to American Society of Anesthesiologist (ASA) class III
* not alert

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2013-12; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Children's Hospital of Eastern Ontario Pain Scale (CHEOPS | up to 1 hour
  The investigators will measure pain scale of sedated children with the CHEOPS (Children's Hospital of Eastern Ontario Pain Scale) during suturing of lacerated wound.

SECONDARY OUTCOMES:
Sedation scale | up to 1 hour
  The investigators will measure sedation scale with Ramsey Sedation Scale.
Complication | up to 1 hour
  The investigators will measure complication with continuous oxygen saturation by pulse oximetry (SpO2) and ECG monitoring and record the monitoring result every 5 minutes.
Satisfaction of parents and clinicians | up to 1 hour
  The investigators will measure Drs. and care givers' satisfaction rate using numeric rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Jin Hee Lee, Professor, Principal Investigator — Seoul National University Bundang Hospital; Jin Hee Lee,, Professor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea